CLINICAL TRIAL: NCT02458898
Title: Text Message Intervention to Improve Adherence in Adolescents and Young Adults With Celiac Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kelly Haas, Principle Investigator, Pediatric Gastroenterology Fellow, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 29967
Record Dates: First submitted 2015-05-21; First posted 2015-06-01 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text Message Intervention (Experimental): A series of 45 unique educational text messages sent over a period of 3 months in the evenings. Text messages include humorous reminders, links to online celiac disease resources, and bidirectional questions.
  Interventions: Behavioral: Educational Text Message Reminders
- Control (No Text Messages) (No Intervention): Routine care by primary gastroenterologist with no text messages.

INTERVENTIONS:
Behavioral: Educational Text Message Reminders — 45 unique text messages designed by the Stanford Pediatric Gastroenterology physicians and nutritionists
  Arms: Text Message Intervention

SUMMARY:
This is a prospective randomized controlled trial investigating the impact of educational bidirectional text message reminders on gluten free diet adherence among adolescents and young adults with celiac disease age 12-24. Participants will complete a series of online questionnaires assessing quality of life, patient activation, celiac symptoms, and self reported dietary adherence at the beginning and end of the study. Participants will also have their blood drawn to measure Tissue Transglutaminase IgA (TTG IgA) antibody and Deamidated Gliadin Peptide IgA (DGP IgA) at the beginning and end of the study. Lab draws can be done locally, and are at no cost to the participant. Patients are randomized to the intervention or control group based on enrollment TTG IgA. Intervention group receives 45 unique text messages over the 3 month study. A gift card is provided for participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-24
* Celiac disease diagnosed by a gastroenterologist at least 1 year prior to enrollment
* Participant with ability to read email and text messages in English
* Access to a mobile phone
* Unlimited text messaging plan or agreement to receive 45 text messages for the study

Exclusion Criteria:

* Participant inability to answer survey questions and text prompts in English

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Tissue Transglutaminase IgA (TTG IgA) | 3 months
  Percent change in TTG IgA for each participant pre and post study period

SECONDARY OUTCOMES:
Deamidated Gliadin Peptide IgA (DGP IgA) | 3 months
  Percent change in DGP IgA for each participant pre and post study period
NIH-PROMIS quality of life score | 3 months
  Change in NIH-PROMIS quality of life questionnaire score pre and post study period
Patient Activation Measure (PAM) score | 3 months
  Change in Patient Activation Measure (PAM) questionnaire score pre and post study period
Patient-reported dietary adherence (CDAT) score | 3 months
  Change in patient-reported dietary adherence (CDAT) questionnaire score pre and post study period
Patient-reported celiac disease symptom measure (CDI) score | 3 months
  Change in patient-reported celiac disease symptom measure (CDI) questionnaire score pre and post study period

CONTACTS AND LOCATIONS:
Overall Officials: Kelly B Haas, MD, Principal Investigator — Stanford Pediatric Gastroenterology
Locations (1):
- Stanford University Pediatric Gastroenterology Department, Palo Alto, California, United States

REFERENCES:
- [Derived] Haas K, Martin A, Park KT. Text Message Intervention (TEACH) Improves Quality of Life and Patient Activation in Celiac Disease: A Randomized Clinical Trial. J Pediatr. 2017 Jun;185:62-67.e2. doi: 10.1016/j.jpeds.2017.02.062. Epub 2017 Mar 23. PMID 28343658
- See also: Study Recruitment Referral Website — https://redcap.stanford.edu/surveys/?s=HYTNWHRAT4